CLINICAL TRIAL: NCT06599424
Title: IntraRenal HEmoDynamics to IntegraTE CA-AKI Risk and Monitor NephroprotectiIoN by ImpElla Support.
Status: Recruiting | Type: Observational
Sponsor: Heinrich-Heine University, Duesseldorf (Other)
Collaborators: German Heart Center (Other); Charite University, Berlin, Germany (Other)
Responsible Party: Sponsor
Other Study IDs: REDETERMINE
Record Dates: First submitted 2024-05-02; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-05

CONDITIONS: Chronic Kidney Diseases; Renal Failure; Coronary Artery Disease
Keywords: CKD; CAD; AKI; nephroprotection; impella; protected PCI
MeSH Terms: conditions — Renal Insufficiency, Chronic; Renal Insufficiency; Coronary Artery Disease | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood and urine samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- subjects with PCI
  Interventions: Other: Observational
- subjectis with Impella-protected PCI
  Interventions: Other: Observational

INTERVENTIONS:
Other: Observational — Observational

SUMMARY:
the hypothesis is that elevation of the intrarenal resistive index (RI) characterizes patients at elevated risk for subsequent CA-AKI and integrates items of the Mehran AKI risk score into a single, readily obtainable parameter. Impella-mediated nephroprotection confers to reduction of elevated RI by restoration of intrarenal venous flow profile.

DETAILED DESCRIPTION:
Contrast-associated acute kidney injury (CA-AKI) occurs in up to 10% of patients undergoing percutaneous coronary intervention (PCI) for coronary revascularization. CA-AKI is associated with impaired long-term outcome. This causes so-called "Renalism", describing the fact that patients with chronic kidney disease (CKD) in need of live-saving revascularizations are not offered PCI procedures in the risk of imminent CA-AKI.

Retrospective studies and one-single-center pilot study described protective effects of Impella-protected PCI to reduce the incidence of CA-AKI. However, mechanisms involved of nephroprotection by Impella remain obscure. Deciphering these, is a prerequisite to tailor nephroprotection to the patients in need and to gain a label for nephroprotection by Impella.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all of the Inclusion Criteria to participate in the trial.

1. Age ≥18 years and <90 years
2. Scheduled for PCI or PROTECTED PCI in near future (1 week) or PCI same day.

Exclusion Criteria:

Subjects must NOT meet any of the following Exclusion Criteria to participate in the trial.

1. Severe chronic kidney disease with eGFR ≤ 20 ml/min or on dialysis
2. Patients with AKI within the last seven days prior screening or incipient AKI (in cases, where AKI cannot be ruled out as a cause for elevated serum creatinine, a rise or fall above 30% of a second serum creatinine measurement obtained within 12 to 24 hours is regarded indicative of AKI).
3. STEMI ≤24 hours from the onset of ischemic symptoms or at any time if mechanical complications of transmural infarction are present (e.g., VSD, papillary muscle rupture, etc.)
4. Cardiogenic shock (SBP <80 mmHg for ≥30 mins and not responsive to intravenous fluids or hemodynamic deterioration for any duration requiring pressors or mechanical circulatory support, including IABP)
5. Cardiorespiratory arrest related to the current admission unless subject is extubated for >24 hours with full neurologic recovery and hemodynamically stable.
6. Platelet count <75,000 cells/mm3, bleeding diathesis or active bleeding, coagulopathy or unwilling to receive blood transfusions.
7. Pregnant or child-bearing potential unless negative pregnancy test within 1 week
8. Participation in the active treatment or follow-up phase of another clinical study of an investigational drug or device that has not reached its primary endpoint
9. Any medical or psychiatric condition such as dementia, alcoholism or substance abuse which may preclude informed consent or interfere with any of the study procedures, including follow-up visits
10. Any non-cardiac condition with life expectancy <1 years (e.g., cirrhosis, cancer not in remission, etc.)
11. Subject belongs to a vulnerable population (defined as individuals with mental disability, persons in nursing homes, impoverished persons, homeless persons, nomads, refugees and those permanently incapable of giving informed consent; vulnerable populations also may include members of a group with a hierarchical structure such as university students, subordinate hospital and laboratory personnel, employees of the Sponsor, members of the armed forces and persons kept in detention)

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with indication for PCI or Impella-protected PCI
Sampling Method: Non-Probability Sample
Enrollment: 550 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-10 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Intrarenal Resistive Index (RI) | immediately and 24 hours after PCI
  unitless, sonographic index measured in intrarenal arteries defined as (peak systolic velocity - end-diastolic velocity ) / peak systolic velocity.
Acute Kidney Injury | 48 hours respectively within 7 days
  Increase in serum creatinine by at least 0.3 mg/dl within 48 hours, or increase in serum creatinine at least 1.5 times the known or assumed baseline value within seven days

SECONDARY OUTCOMES:
Serum creatinine (mg/dl) and calculated creatinine clearance (ml/min) in relation to RI (Intrarenal Resistive Index) an Mehran score (unitiles) | maximum change 24 hours post intervention compared to baseline
  Relation calculated by Pearson correlation
α2macroglobulin urine concentration in relation to RI and Mehran score (unitiless). | maximum change 24 hours post intervention compared to baseline
  Relation calculated by Pearson correlation
NGAL urine concentration (ng/ml) in subgroup analysis in relation to RI and mehran score (unitless); | maximum change 24 hours post intervention compared to baseline
  Relation calculated by Pearson correlation
Reclassification of AKI Risk by determined cutoff value for RI compared to classic Mehran score | maximum change day 1 or day 2 post intervention compared to baseline
Length of stay in relation to RI and classic Mehran score. | Hospital admission until discharge (assessed up to maximum of 10 days)
Hierarchical clinical endpoint of AKI > rise of urinary α2macroglobulin concentration post PCI > increase of RI post PCI in Impella-protected patients versus non-Impella-protected patients matched by Mehran score | maximum change day 1 or day 2 post intervention compared to baseline
Change of RI (Intrarenal Resistive Index) by Impella comparing RI at performance levels P0 and P9 at the begin of the intervention in every Impella-protected patient. | during Impella treatment (up to 14 days)

CONTACTS AND LOCATIONS:
Overall Officials: Malte Kelm, Prof., Study Chair — Division of Cardiology, Pulmonary Disease and Vascular Medicine; Amin Polzin, Prof., Principal Investigator — Division of Cardiology, Pulmonary Disease and Vascular Medicine
Locations (2):
- Germany (2):
  - Department of Cardiology, Angiology and Intensive Care Medicine Campus at German Heart Center Charite, Berlin
  - Division of Cardiology, Pulmonary Disease and Vascular Medicine at University Hospital Duesseldorf, Düsseldorf

IPD SHARING:
Plan to Share IPD: No